CLINICAL TRIAL: NCT05977153
Title: CT-Guided Personalized Mechanical Ventilation to Minimize Ventilator-Induced Lung Injury Study
Brief Title: CT for Personalized Mechanical Ventilation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Charles W. Emala, Henrik H. Bendixen Professor of Anesthesiology, Vice Chair of Research in the Department of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT8623; 5R01HL121228-09 (NIH)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Ventilator-Induced Lung Injury; Sepsis Syndrome; Mechanical Ventilation Complication
Keywords: Computed Tomography; Registration Analysis; Functional Lung Imaging; Acute Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Systemic Inflammatory Response Syndrome; Acute Lung Injury | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ARDSNet (Active Comparator): Participants will receive standard ARDSNet low-stretch PEEP (positive end-expiratory pressure) protocol.
  Interventions: Procedure: PEEP (positive end-expiratory pressure) - standard
- Group 2: Individualized PEEP (positive end expiratory pressure) Strategy (Experimental): Participants will receive individualized PEEP (positive end-expiratory pressure).
  Interventions: Procedure: PEEP (positive end-expiratory pressure) - maximum

INTERVENTIONS:
Procedure: PEEP (positive end-expiratory pressure) - maximum — Breathing assistance from the breathing assist machine using a method in which doctors try to find the pressures that expands the lungs the best. This is based on measurements of one's respiratory pressures and volumes. This is done by adjusting the pressure settings. This allows one's lungs to expand with the least amount of change in pressure during breathing.
  PEEP (positive end-expiratory pressure) will be set at the maximum static respiratory system compliance (Crs) during a descending PEEP titration curve.
  Arms: Group 2: Individualized PEEP (positive end expiratory pressure) Strategy
Procedure: PEEP (positive end-expiratory pressure) - standard — Breathing assistance from the breathing assist machine using the pressure settings typical for your disease.
  Standard ARDSNet low-stretch PEEP (positive end-expiratory pressure) protocol: PEEP will be set following a routinely used PEEP table according to patients' blood oxygenation status.
  Arms: Group 1: ARDSNet

SUMMARY:
The goal of this study is to compare two different ways of helping patients with a condition called sepsis who need help breathing using a machine called a ventilator. The investigators want to study which way of setting the ventilator is better for the lungs.

Here are the main questions the investigators want to answer:

1. How does the amount of air in the lungs and the way it moves differ between the two ways?
2. How does the way air spreads out in different parts of the lungs differ between the two ways? In this study, the investigators will take special pictures of the lungs using a machine called a CT scan. The pictures will show us how much the lungs stretch and how much air is in different parts of the lungs. The investigators will compare two different ways of using the ventilator: one personalized for each patient based on their breathing, and another way that is commonly used.

By comparing these two ways, the investigators hope to learn which one is better for helping patients with sepsis who need the ventilator. This information can help doctors make better decisions about how to care for these patients and improve their breathing.

DETAILED DESCRIPTION:
Mechanical ventilation is a key life support method applied to millions of surgical and critically ill patients. Ventilator-induced lung injury (VILI) is a major factor for morbidity and mortality in patients with the acute respiratory distress syndrome (ARDS), the most severe form of respiratory dysfunction. Furthermore, mechanical ventilation settings also contribute to the risk for postoperative pulmonary complications (PPCs) in surgical patients and lung injury in critically ill patients with normal lungs at onset of ventilation. In summary, mitigation of VILI is critical to reduce perioperative and critical care morbidity and mortality, with major impact on outcomes and health care costs.

In this project, we propose to apply novel CT methods to assess spatial distributions of strain and aeration and establish measures of global lung mechanics best indicative of the PEEP leading to least injurious distributions and, thus, least VILI.

ELIGIBILITY:
Inclusion Criteria:

* Following onset of mechanical ventilation and not longer than 5 days after intubation.
* Sepsis as defined by the most recent criteria:

  * Life-threatening organ dysfunction caused by a dysregulated host response to infection operationalized by presumed or documented infection and a Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score >= 2 or a change by 2 from the baseline if baseline known to be different from 0;

Exclusion Criteria:

* Age < 18 years;
* Hemodynamic instability, defined as: systolic blood pressure (SBP) < 90 mmHg that is not adequately stabilized by vasopressors or inotropic agents. For these purposes, SBP will not be considered "adequately stabilized" if the dose of the vasopressor/inotrope has not been stable for at least one hour;
* Hypoxemia, defined as: PaO2 < 70 mmHg on an inspired oxygen fraction (FiO2) greater than or equal to 0.9;
* Hemodynamic and/or respiratory instability (as defined, in items 2 and 3) that develop when the patient is mobilized during routine nursing care such as repositioning/washing the patient or changing their bed linens;
* Hemodynamic and/or respiratory instability (as defined, in items 2 and 3) that develop when a 20 second respiratory pause is required to implement the study protocol. This will be tested by inducing such a pause prior to transporting the patient;
* Any acute or chronic condition which, in the opinion of the investigators, might confound the imaging measurements (such as, but not limited to, severe bronchospasm, pulmonary infection, and lung tumor);
* Any acute or chronic condition which, in the opinion of the investigators or managing critical care team, could prevent safe transport to the CT suite.
* "Air leaks" requiring tube thoracotomy (e.g., pneumothorax, bronchopleural fistula);
* Body mass index > 40 kg/m2;
* Pregnancy (since this is a study that would expose a fetus to radiation risk);
* Patients who have taken part in other research studies involving radiation exposure, or those patients for whom this research radiation history is unavailable at the time of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Squared coefficient of variation of the tidal volumetric strain | 48 hours
  Squared coefficient of variation (=variance normalized by the squared mean) of the tidal volumetric strain will be obtained and calculated from CT images.

SECONDARY OUTCOMES:
Squared coefficient of variation of aeration | 48 hours
  Squared coefficient of variation (=variance normalized by the squared mean) of aeration obtained and calculated from CT images.
Average gas fraction | 48 hours
  Average gas fraction will be obtained and calculated from CT images.
Distribution of aeration categories | 48 hours
  Distribution of aeration categories (non-aerated, poorly aerated, normally aerated and hyperinflated regions) will be obtained and calculated from CT images.
Average tidal strain | 48 hours
  Average of voxel level volumetric tidal strain will be obtained and calculated from CT images.

OTHER OUTCOMES:
Time during mechanical ventilation | Up to 5 days
  Time during mechanical ventilation will be recorded in days.
Detection of Inflammatory cytokines | 48 hours
  Inflammatory cytokine is a type of signaling molecule (a cytokine) that is secreted from immune cells like helper T cells (Th) and macrophages, and certain other cell types that promote inflammation; their presence will be measured by assays.

CONTACTS AND LOCATIONS:
Overall Officials: Charles W. Emala, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a NIH funded study. Data sharing will follow NIH guidelines.